CLINICAL TRIAL: NCT04730245
Title: Targeting Gut Microbiota for Motor Complications in Parkinson´s Disease
Brief Title: Microbiota Modification for the Treatment of Motor Complication of Parkinson´s Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torre Médica Santé (Network)
Responsible Party: Principal Investigator, José Fidel Baizabal-Carvallo, Neurologist, physician, investigator, Torre Médica Santé
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202004-001
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease Aggravated
Keywords: Parkinson´s disease; Constipation; Dyskinesia; Microbiota
MeSH Terms: conditions — Parkinson Disease; Constipation; Dyskinesias | interventions — Rifaximin; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microbiota modification (Experimental)
  Interventions: Drug: sodium phosphate enema, oral rifaximin and polyethylene glycol

INTERVENTIONS:
Drug: sodium phosphate enema, oral rifaximin and polyethylene glycol — Patients were hospitalized for 4-5 hours to receive two saline colon enemas with sodium phosphate Fleet®, 2 to 3 hours apart, appropriate hydration was provided during the procedure. If signs of fecal impaction were observed, the stools were removed manually prior to the first enema. Patients were discharged with oral treatment consistent with rifaximin 200 mg three times a day for 7 days and polyethylene glycol-3350, 17 gr per day in water for 10 days, but it was continued if necessary. Importantly, no modifications in time and dose of dopaminergic therapy or anti-dyskinetic medication (i.e. amantadine) were done at baseline or during the study

SUMMARY:
In recent years, abnormalities in gut microbiota have been identified in patients with Parkinson´s disease having a possible role in motor manifestations. Among 80 patients with PD, we selected 14 with LID and motor fluctuations with limited response to pharmacological therapy to receive treatment with sodium phosphate enema, oral rifaximin and polyethylene glycol to improve motor complications.

DETAILED DESCRIPTION:
We studied consecutive patients diagnosed with PD according to the Queen Square Brain Bank Criteria [Hughes et al 1992] in a tertiary care center for movement disorders, from June 2018 to March 2020.

ELIGIBILITY:
Inclusion Criteria:

- patients aged 18-years old or older with moderate to severe dyskinesia and/or motor fluctuations with incomplete or poor response to adjustments in time and dose of levodopa and other anti-parkinsonian agents such as entacapone, rasagiline, dopamine receptor agonists and amantadine in 1-2 months prior to enrollment; defined by a Movement Disorders Society Unified Parkinson´s Disease Rating Scale (MDS-UPDRS) part IV score equal or higher than 8 following pharmacological adjustments.

Exclusion Criteria:

* patients with chronic renal failure, decompensated heart failure, colonic abnormalities precluding the use of evacuating enema, known allergies to prescribed medications to reduce microbiota load and patients who declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Improvement in MDS-UPDRS-IV score | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: José Fidel Baizabal-Carvallo, M.D., Principal Investigator — Torre Médica Sante
Locations (1):
- Torre Medica Sante, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
May be shared by specific request